CLINICAL TRIAL: NCT00232609
Title: Development of the GameCycle Exercise System: Phase II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Rory Cooper, PhD, Human Engineering Research Laboratories
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 02254, 0410155; 2R44HD039535-02A1 (NIH)
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Wheelchair Users
Keywords: Wheelchair; Exercise; Cardiovascular Disease
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GameCycle Exercise System

SUMMARY:
The purpose of this research project is to further develop and test the effectiveness of a novel exercise system for wheelchair users, the Game Cycle.

DETAILED DESCRIPTION:
The purpose of this research project is to further develop and test the effectiveness of a novel exercise system for wheelchair users, the GAMECycle. People in wheelchairs who have a desire to exercise are faced with barriers with respect to access to exercise equipment and to availability of exercise equipment that is specifically suitable for use with a wheelchair. The GAMECycle exercise system removes these barriers and offers the wheelchair user an entertaining, motivational environment in which to exercise. The long-term goal is to improve the overall activity level of individuals who use wheelchairs as their primary means of mobility and increase their general well being.

The GAMECycle Exercise System is a modified arm-ergometer that sits on a turnstile to allow steering in much the same way as an arm-cycle. More specifically, it is a crank and pedal set that is turned using the arms, similar to a bicycle that is turned with the feet. When using the system, subjects will be seated in their own wheelchair in front of the system comfortably positioned to be able to grasp the handles and use the arm crank. The GAMECycle is designed to provide upper body aerobic exercise in an environment (computer game play) that will help to make exercise more enjoyable by, among other things, distracting people from some of the less pleasant aspects of exercising. Although upper-body exercise systems for wheelchair users do exist, the GAMECycle is unique in its ability to combine arm-ergometry with playing computer videogames. And, in contrast to wheelchair roller systems, the arm-ergometry provided by the GAMECycle affords the user an exercise option that uses a motion that differs significantly from the motion of wheelchair propulsion.

This research consists of two phases: a Training Phase and an In Home Trial Phase. The training phase will last a maximum of two hours and the In Home Phase will last 4 months. Subjects who complete the Training Phase will be asked to participate in the In Home Trial.

Training Phase The purpose of the training sessions are to determine the users ability to reach and maintain target aerobic training zones during 15 minute exercise trials, teach new users how to use the GAMECycle Exercise System, and to obtain feedback from new users regarding perceived comfort, fit, and ease of use.

A GAMECycle exercise system will be set up in participating local rehab and research facilities. A clinician will ensure that the GAMECycle is adjusted to fit each user. The amount of resistance from the arm-ergometer will be adjusted to a level that feels comfortable during exercise. Heart rate and breathing rate will be monitored during a 15-minute exercise session. Subjects will rate their level of exertion every 2 minutes during the 15-minute exercise phase and will be asked to complete a questionnaire about their opinion of the GAMECycle System.

In Home Phase This phase involves a 4-month trial period divided into 2 two-month sessions. For two months, subjects will be asked to use the GAMECycle and for the other two months, subjects will be asked to use an arm-ergometer. It will randomly be determined whether the GAMECycle or the arm-ergometer is used first. Subjects will be required to record their exercise sessions and will be followed by a member of the research team by telephone. In addition, once a month for four months, a member of our research staff will visit each participant with a portable metabolic cart and heart rate monitor in order to collect heart rate date, metabolic date (VO2, VCO2), and ratings of perceived exertion using the Borg scale. This data will be collected during exercise with or without game play, depending on the condition of that session.

ELIGIBILITY:
Inclusion Criteria:

1. Use of a wheelchair as primary means of mobility (use a wheelchair > 20 hours per week)
2. Between ages 18 and 50
3. Able to use an arm-cycle

Exclusion Criteria:

1. Any history of cardiovascular or cardiopulmonary disease for the participant, or a history of CVD in their family (e.g., parents, grandparents, and siblings) which will be defined as death as a result of CVD prior to the age of 55.
2. If a subject answers yes to any question on the PAR-Q.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2005-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Physiologic and Metabolic activity (VO2, VCO2, HR)
Ratings of perceived exertion
Questionnaire responses

CONTACTS AND LOCATIONS:
Overall Officials: Rory A Cooper, PhD, Principal Investigator — University of Pittsburgh and VA Pittsburgh Healthcare System
Locations (1):
- Human Engineering Research Laboratories, Pittsburgh, Pennsylvania, United States